CLINICAL TRIAL: NCT03489720
Title: Evaluation of a Daily Brief Exercise Intervention on Resident Physician Personal Resiliency and Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Uma Shastri, Assistant Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 180313
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-02

CONDITIONS: Burnout, Professional; Burnout Syndrome
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: balanced order-randomized, 16-week within-subject crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Exercise intervention then usual exercise program (Experimental): 8 weeks of exercise intervention followed by 8 weeks of usual exercise program
  Interventions: Behavioral: Prescribed Exercise Program; Behavioral: Usual Exercise Program
- Arm B: Usual Exercise Program then exercise intervention (Active Comparator): 8 weeks of usual exercise program followed by 8 weeks of exercise intervention
  Interventions: Behavioral: Prescribed Exercise Program; Behavioral: Usual Exercise Program

INTERVENTIONS:
Behavioral: Prescribed Exercise Program — Brief cardiovascular exercise training (>70% of maximum heart rate) for 15 minutes a day, 5 days a week for 8 weeks.
  The exercise intervention will be a 15-minute per day of vigorous exercise that as monitored by a Fitbit Charge 2.
  Examples of possible 15-minute exercise regimens to be used include:
  * Walking quickly or running up and down stairs
  * Plyometric exercises such as jumping jacks, high knees, squats, lunges, speed skaters, froggers, etc
  * Walking up an incline on a treadmill
  * Jogging or running on a treadmill or elliptical
  * Stationary cycling or rowing
Behavioral: Usual Exercise Program — Usual exercise activity for 8 weeks

SUMMARY:
This study seeks to evaluate the prevalence and characterize predictors of physician burnout in the anesthesia residency at Vanderbilt University Medical Center. The study also seeks to evaluate the effect of an exercise intervention on burnout and personal resiliency (i.e., less individual stress given the same workload).

DETAILED DESCRIPTION:
A cross-sectional evaluation of burnout, perceived stress, average sleep propensity, and social support and coping mechanisms will be assessed from four years of Vanderbilt University Medical Center (VUMC) Anesthesia residents. Burnout will be assessed using the Maslach Burnout Inventory (MBI-HSS).

Participating interns, Anesthesia Residency Class 1 (CA-1), and Anesthesia Residency Class 2 (CA-2) classes will be randomized to 8 weeks of an exercise intervention (15 min of activity at 70% of max heart rate or higher, 5 days a week) to meet the activity recommendations of the Office of Disease Prevention and Health Promotion or 8 weeks of continuing their baseline activity level prior to the study.

ELIGIBILITY:
Inclusion Criteria:

* Vanderbilt University Medical Center Anesthesiology residents (Class 1(CA-1), Class 2 (CA-2)

Exclusion Criteria:

* Failure to sign informed consent
* Will not be in town and available for the full duration of the study (e.g., 2 or more weeks of vacation or absence)
* Physical inability to perform the exercise intervention (including health indications)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uma Shastri, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Unversity Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were randomized to intervention arm followed by control arm. These participants withdrew from the study after the start of the intervention arm and never started the control arm.
Period: Overall Study
Arm/Group | Arm A: Exercise Intervention Then Usual Exercise Program | Arm B: Usual Exercise Program Then Exercise Intervention
Started | 24 | 22
Completed | 22 | 22
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exercise Intervention Then Usual Exercise Program: 8 weeks of exercise intervention followed by 8 weeks of usual exercise program
- Usual Exercise Program Then Exercise Intervention: 8 weeks of usual exercise program followed by 8 weeks of exercise intervention
- Total: Total of all reporting groups
Arm/Group | Exercise Intervention Then Usual Exercise Program | Usual Exercise Program Then Exercise Intervention | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 46
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 10 | 10 | 20
  Not reported | 3 | 0 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Emotional Exhaustion (EE) Burnout Score(as Measured by the Maslach Burnout Inventory (MBI)From Baseline to End of Each Exercise Phase.
Description: The change in the Emotional Exhaustion (EE) burnout score(as measured by the Maslach Burnout Inventory (MBI)from baseline to end of each exercise phase.
  MBI-HSS is a survey to measure burnout in professionals in human services. MBI-HSS EE score includes 9 items to evaluate emotional exhaustion (EE), with scores ranging from 0 to 6 on the Likert scale. MBI-HSS EE total score ranges from 0 to 54 points. We consider a high degree of burnout in the case of EE ≥ 27 points. Moderate burnout will be considered in the case of 26<EE<19 points. Low levels will be considered for EE≤18 points.
Time Frame: Baseline to 8 weeks
Population: Data was not available for analysis of baseline data for 1 participant in each exercise phase.
  Data was not available for analysis of change in MBI-EE for 2 participants in each exercise phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Exercise Intervention: Prescribed Exercise Program: Brief cardiovascular exercise training (>70% of maximum heart rate) for 15 minutes a day, 5 days a week for 8 weeks.
  The exercise intervention will be a 15-minute per day of vigorous exercise that as monitored by a Fitbit Charge 2.
  Examples of possible 15-minute exercise regimens to be used include:
  * Walking quickly or running up and down stairs
  * Plyometric exercises such as jumping jacks, high knees, squats, lunges, speed skaters, froggers, etc
  * Walking up an incline on a treadmill
  * Jogging or running on a treadmill or elliptical
  * Stationary cycling or rowing
  Usual Exercise Program: Usual exercise activity for 8 weeks
Arm/Group | Exercise Intervention | Usual Exercise Program
Number analyzed (Participants) | 44 | 44
units on a scale
  Baseline: number analyzed (Participants) | 43 | 43
  Baseline | 20.95348837 (9.756447168) | 20.93023256 (10.40694674)
  Change after 8 weeks of exercise phase: number analyzed (Participants) | 42 | 42
  Change after 8 weeks of exercise phase | -0.976190476 (7.416159335) | -0.095238095 (6.472491599)

2. Primary Outcome: The Change in the Depersonalization (DP) Burnout Score(as Measured by the Maslach Burnout Inventory (MBI))From Baseline to End of Each Exercise Phase.
Description: The change in the Depersonalization (DP) burnout score(as measured by the Maslach Burnout Inventory (MBI))from baseline to end of each exercise phase.
  MBI-HSS is a survey to measure burnout in professionals in human services. MBI-HSS DP score includes 5 items to evaluate depersonalization (DP) with scores ranging from 0 to 6 on the Likert scale. MBI-HSS DP total score ranges from 0 to 30 points. We consider a high degree of burnout in the case of DP≥ 13 points. Moderate burnout will be considered in the case of 7-12 DP points. Low levels will be considered for DP ≤6 points.
Time Frame: Baseline to 8 weeks
Population: Data was not available to analyze the change from baseline in one participant for the exercise intervention period.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Exercise Intervention: Prescribed Exercise Program: Brief cardiovascular exercise training (>70% of maximum heart rate) for 15 minutes a day, 5 days a week for 8 weeks.
  The exercise intervention will be a 15-minute per day of vigorous exercise that as monitored by a Fitbit Charge 2.
  Examples of possible 15-minute exercise regimens to be used include:
  * Walking quickly or running up and down stairs
  * Plyometric exercises such as jumping jacks, high knees, squats, lunges, speed skaters, froggers, etc
  * Walking up an incline on a treadmill
  * Jogging or running on a treadmill or elliptical
  * Stationary cycling or rowing
Arm/Group | Exercise Intervention | Usual Exercise Program
Number analyzed (Participants) | 43 | 43
units on a scale
  Baseline | 8.465116279 (4.762696501) | 8.181818182 (5.077413402)
  Change after 8 weeks of usual exercise program: number analyzed (Participants) | 42 | 43
  Change after 8 weeks of usual exercise program | 0.139534884 (3.412731034) | -0.727272727 (3.743916842)

3. Primary Outcome: The Change in the Personal Accomplishment (PA) Burnout Score(as Measured by the Maslach Burnout Inventory (MBI))From Baseline to End of Each Exercise Phase.
Description: The change in the Personal Accomplishment (PA) burnout score(as measured by the Maslach Burnout Inventory (MBI))from baseline to end of each exercise phase.
  MBI-HSS is a survey to measure burnout in professionals in human services. MBI-HSS PA score includes 8 items to evaluate Personal Accomplishment (PA) with scores ranging from 0 to 6 on the Likert scale. MBI-HSS PA total score ranges from 0 to 48 points. We consider a high degree of burnout in the case of PA≥ 39 points. Moderate burnout will be considered in the case of 32-38 PA points. Low levels will be considered for PA ≤31 points.
Time Frame: Baseline to 8 weeks
Population: Data was available for analysis of change for 43 (exercise intervention) and 42 (usual exercise)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Intervention | Usual Exercise Program
Number analyzed (Participants) | 44 | 43
units on a scale
  Baseline | 34.13636364 (6.729286596) | 34.95348837 (7.107854436)
  Change after 8 weeks of usual exercise program: number analyzed (Participants) | 43 | 42
  Change after 8 weeks of usual exercise program | 0.209302326 (6.235681272) | 0.738095238 (5.355915461)

4. Primary Outcome: Change in the Emotional Exhaustion (EE) Burnout Score(as Measured by MBI From Baseline to End of Each Exercise Phase Stratified by Training Level (Post Graduate Year 1 (PGY1), Post Graduate Year 2 (PGY2), and Post Graduate Year 3 (PGY3))
Description: The change in the Emotional Exhaustion burnout score(as measured by the Maslach Burnout Inventory (MBI)from baseline to end of each exercise phase stratified by training level.
  MBI-HSS is a survey to measure burnout in professionals in human services. MBI-HSS includes 9 items to evaluate emotional exhaustion (EE) with scores ranging from 0 to 6 on the Likert scale. MBI-HSS EE total score ranges from 0 to 54 points. We consider a high degree of burnout in the case of EE ≥ 27 points. Moderate burnout will be considered in the case of 26<EE<19 points. Low levels will be considered for EE≤18 points.
Time Frame: Baseline to 8 weeks
Population: 16 PGY1, 13 PGY2, &15 PGY3 participated in study. Data not available in 1 PGY1 participant in exercise intervention period. Data not available to assess change after usual exercise period for 1 PGY2 participant. Data not available for 1 PGY3 participnt for baseline or change in usual exercise period, & change in 1 participant exercise intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Intervention | Usual Exercise Program
Number analyzed (Participants) | 44 | 44
units on a scale
  Post graduate year 1: Baseline: number analyzed (Participants) | 15 | 16
  Post graduate year 1: Baseline | 21.2 (10.37992568) | 20.125 (11.43022309)
  Post graduate year 1: Change after 8 weeks: number analyzed (Participants) | 15 | 16
  Post graduate year 1: Change after 8 weeks | -2.266666667 (5.66274374) | -2.0625 (6.287222492)
  Post graduate year 2: Baseline: number analyzed (Participants) | 13 | 13
  Post graduate year 2: Baseline | 20.84615385 (9.948585778) | 20.84615385 (10.07344822)
  Post graduate year 2: Change after 8 weeks: number analyzed (Participants) | 12 | 13
  Post graduate year 2: Change after 8 weeks | 1.846153846 (8.434513954) | 0.833333333 (5.89067059)
  Post graduate year 3: Baseline: number analyzed (Participants) | 15 | 14
  Post graduate year 3: Baseline | 20.8 (9.637723501) | 21.92857143 (10.17889435)
  Post graduate year 3: Change after 8 weeks: number analyzed (Participants) | 14 | 14
  Post graduate year 3: Change after 8 weeks | -2.214285714 (7.856193749) | 2.071428571 (6.521730371)

5. Primary Outcome: The Change in the Depersonalization (DP) Burnout Score(as Measured by the Maslach Burnout Inventory (MBI))From Baseline to End of Each Exercise Phase Stratified by Training Level.
Description: The change in the Depersonalization (DP) burnout score(as measured by the Maslach Burnout Inventory (MBI))from baseline to end of each exercise phase stratified by training level.
  MBI-HSS is a survey to measure burnout in professionals in human services. DP MBI-HSS includes 5 items to evaluate depersonalization (DP) with scores ranging from 0 to 6 on the Likert scale. MBI-HSS DP total score ranges from 0 to 30 points. We consider a high degree of burnout in the case of DP ≥ 10. Moderate burnout will be considered in the case of 6<DP<9 points. Low levels will be considered for DP≤5 points.
Time Frame: Baseline to 8 weeks
Population: There were 16 PGY1, 13 PGY2, and 15 PGY3 participants in study. Data available in 15 PGY1 participants in exercise intervention period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Intervention | Usual Exercise Program
Number analyzed (Participants) | 44 | 44
units on a scale
  Post graduate year 1: Baseline: number analyzed (Participants) | 15 | 16
  Post graduate year 1: Baseline | 6.866666667 (4.596064569) | 6.3125 (5.055937104)
  Post graduate year 1: Change after 8 weeks: number analyzed (Participants) | 15 | 16
  Post graduate year 1: Change after 8 weeks | -1.266666667 (2.865226659) | -1.8125 (4.354595274)
  Post graduate year 2: Baseline: number analyzed (Participants) | 13 | 13
  Post graduate year 2: Baseline | 9.461538462 (4.502136245) | 9.615384615 (4.233565509)
  Post graduate year 2: Change after 8 weeks: number analyzed (Participants) | 13 | 13
  Post graduate year 2: Change after 8 weeks | 0.846153846 (3.262058497) | -0.076923077 (2.985005261)
  Post graduate year 3: Baseline: number analyzed (Participants) | 15 | 15
  Post graduate year 3: Baseline | 9.2 (5.031330412) | 8.933333333 (5.470265946)
  Post graduate year 3: Change after 8 weeks: number analyzed (Participants) | 15 | 15
  Post graduate year 3: Change after 8 weeks | 0.933333333 (3.788453636) | 0.4 (3.581699517)

6. Primary Outcome: The Change in the Personal Accomplishment (PA) Burnout Score(as Measured by the Maslach Burnout Inventory (MBI))From Baseline to End of Each Exercise Phase Stratified by Training Level.
Description: The change in the PA burnout score(as measured by the Maslach Burnout Inventory (MBI))from baseline to end of each exercise phase stratified by training level.
  MBI-HSS is a survey to measure burnout in professionals in human services. PA MBI-HSS includes 8 items to evaluate personal accomplishment (PA), with scores ranging from 0 to 6 on the Likert scale. MBI-HSS PA total score ranges from 0 to 48 points. We consider a high degree of burnout in the case of PA≥ 39 points. Moderate burnout will be considered in the case of 32-38 PA points. Low levels will be considered for PA ≤31 points.
Time Frame: Baseline to 8 weeks
Population: There were 16 PGY1, 13 PGY2, and 15 PGY3 participants in study. Data available in 15 PGY1 participants for change in exercise intervention period and baseline in usual exercise period, and change in 13 participants after usual exercise program.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Intervention | Usual Exercise Program
Number analyzed (Participants) | 44 | 43
units on a scale
  Post graduate year 1: Baseline: number analyzed (Participants) | 16 | 15
  Post graduate year 1: Baseline | 33 (7.456540753) | 34.2 (7.775419144)
  Post graduate year 1: Change after 8 weeks: number analyzed (Participants) | 15 | 13
  Post graduate year 1: Change after 8 weeks | -0.2 (6.635402884) | 1.428571429 (5.243520334)
  Post graduate year 2: Baseline: number analyzed (Participants) | 13 | 13
  Post graduate year 2: Baseline | 36.15384615 (6.2695847) | 36.38461538 (6.776656766)
  Post graduate year 2: Change after 8 weeks: number analyzed (Participants) | 13 | 13
  Post graduate year 2: Change after 8 weeks | 1 (4.795831523) | 1 (5.016638981)
  Post graduate year 3: Baseline: number analyzed (Participants) | 15 | 15
  Post graduate year 3: Baseline | 33.6 (6.344851681) | 34.46666667 (6.998639324)
  Post graduate year 3: Change after 8 weeks: number analyzed (Participants) | 15 | 15
  Post graduate year 3: Change after 8 weeks | 0.466666667 (7.199867724) | -0.133333333 (5.962581735)

7. Primary Outcome: The Degree of Burnout Among VUMC Anesthesia Interns and Residents as Quantified by Baseline Emotional Exhaustion (EE) MBI-HSS Scores Broken Down by Level of Residency Training Completed.
Description: The degree of burnout among VUMC anesthesia interns and residents as quantified by baseline Emotional Exhaustion MBI-HSS scores broken down by level of residency training completed.
  MBI-HSS is a survey to measure burnout in professionals in human services. MBI-HSS EE score includes 9 items to evaluate emotional exhaustion (EE), with scores ranging from 0 to 6 on the Likert scale. MBI-HSS EE total score ranges from 0 to 54 points. We consider a high degree of burnout in the case of EE ≥ 27 points. Moderate burnout will be considered in the case of 26<EE<19 points. Low levels will be considered for EE≤18 points.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Post Graduate Year 1: VUMC anesthesia post medical school graduate year 1
- Post Graduate Year 2: VUMC anesthesia post medical school graduate year 2
- Post Graduate Year 3: VUMC anesthesia post medical school graduate year 3
Arm/Group | Post Graduate Year 1 | Post Graduate Year 2 | Post Graduate Year 3
Number analyzed (Participants) | 17 | 15 | 14
units on a scale | 20.29412 (8.858363) | 16.80000 (10.255312) | 27.64286 (12.481415)

8. Primary Outcome: The Degree of Burnout Among VUMC Anesthesia Interns and Residents as Quantified by Baseline Depersonalization MBI-HSS Scores Broken Down by Level of Residency Training Completed.
Description: The degree of burnout among VUMC anesthesia interns and residents as quantified by baseline Depersonalization MBI-HSS scores broken down by level of residency training completed.
  MBI-HSS is a survey to measure burnout in professionals in human services. MBI-HSS DP score includes 5 items to evaluate depersonalization (DP) with scores ranging from 0 to 6 on the Likert scale. MBI-HSS DP total score ranges from 0 to 30 points. We consider a high degree of burnout in the case of DP≥ 13 points. Moderate burnout will be considered in the case of 7-12 DP points. Low levels will be considered for DP ≤6 points.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post Graduate Year 1 | Post Graduate Year 2 | Post Graduate Year 3
Number analyzed (Participants) | 17 | 15 | 14
units on a scale | 7.647059 (5.086025) | 6.266667 (4.817626) | 9.357143 (6.570413)

9. Primary Outcome: The Degree of Burnout Among VUMC Anesthesia Interns and Residents as Quantified by Baseline Personal Accomplishment (PA) MBI-HSS Scores Broken Down by Level of Residency Training Completed.
Description: The degree of burnout among VUMC anesthesia interns and residents as quantified by baseline Personal Accomplishment MBI-HSS scores broken down by level of residency training completed.
  MBI-HSS is a survey to measure burnout in professionals in human services. MBI-HSS PA score includes 8 items to evaluate Personal Accomplishment (PA) with scores ranging from 0 to 6 on the Likert scale. MBI-HSS PA total score ranges from 0 to 48 points. We consider a high degree of burnout in the case of PA≥ 39 points. Moderate burnout will be considered in the case of 32-38 DP points. Low levels will be considered for DP ≤31 points.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post Graduate Year 1 | Post Graduate Year 2 | Post Graduate Year 3
Number analyzed (Participants) | 17 | 15 | 14
units on a scale | 34.41176 (6.828788) | 34.60000 (8.584038) | 33.35714 (9.352969)

ADVERSE EVENTS:
Time Frame: 16 weeks of study participation
Arm/Group | Exercise Intervention | Usual Exercise Program
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 0/46 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT03489720/Prot_SAP_000.pdf